CLINICAL TRIAL: NCT06609759
Title: Efficacy and Safety of Postoperative Adjuvant Therapy for Stage II-III Gastric Cancer: a Prospective, Observational Study
Brief Title: Postoperative Adjuvant Therapy for Stage II-III Gastric Cancer
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Jinan Central Hospital (Other); Yantai Yuhuangding Hospital (Other); The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Lian Liu, MD, PHD, Professor, Chief Physician, Qilu Hospital of Shandong University
Other Study IDs: MRD2
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Stage II-III Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard chemotherapy regimen
  Interventions: Drug: Standard chemotherapy regimen

INTERVENTIONS:
Drug: Standard chemotherapy regimen — In terms of postoperative adjuvant treatment, treatment is based on the guideline standard treatment plan, which can be adjusted according to the doctor's experience.

SUMMARY:
For patients with stage II-III gastric cancer after radical D2 resection and R0 resection, postoperative adjuvant therapy guided by ctDNA-MRD (MRD-GATE external cohort) was not inferior to the standard chemotherapy regimen (this cohort).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone D2 gastrectomy, achieved R0 resection, and are pathologically diagnosed with stage II-III gastric cancer.
2. No preoperative neoadjuvant or adjuvant therapy received.
3. Voluntary participation with signed informed consent, demonstrating good compliance and willingness to cooperate with follow-up procedures.
4. Age between 18-75 years, with no gender restrictions.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Estimated survival of 6 months or more.
7. Baseline hematological and biochemical parameters within specified limits: a. Hemoglobin ≥ 80g/L. b. Absolute neutrophil count ≥ 1.5×10^9/L. c. Platelet count ≥ 100×10^9/L. d. Aspartate or alanine aminotransferase ≤ 2.5 times the upper limit of normal. e. Alkaline phosphatase ≤ 2.5 times the upper limit of normal. f. Thyroid-stimulating hormone (TSH) ≤ 1 times the upper limit of normal (if abnormal, T3 and T4 levels must be normal).

Exclusion Criteria:

1. Pregnant or lactating women, or women of childbearing potential with a positive pregnancy test at baseline.
2. Evidence of postoperative recurrence or metastasis.
3. Previous anti-tumor therapy, including chemotherapy, radiotherapy, or immunotherapy.
4. Positive resection margins identified in postoperative pathology.
5. History of other malignancies within the past five years, except certain skin cancers, superficial bladder cancer, in situ cervical or breast cancer.
6. Uncontrolled pleural effusion, pericardial effusion, or ascites.
7. Severe cardiovascular conditions such as symptomatic coronary artery disease, congestive heart failure (grade ≥ II), uncontrolled arrhythmias, or myocardial infarction within the last 12 months.
8. Uncontrolled infection, severe kidney disease, or other significant concurrent diseases.
9. Allergic reactions to study drugs.
10. Receipt of any anti-tumor therapy within 4 weeks prior to enrollment.
11. Administration of live attenuated vaccines within 4 weeks prior to the first study treatment dose or plans to receive such vaccines during the study period.
12. Positive HIV antibody, active hepatitis B or C (with specific viral load criteria).
13. Positive for COVID-19 nucleic acid or antigen test.
14. Other conditions deemed by the investigator to potentially affect patient safety or trial compliance, including serious illnesses requiring treatment, severe laboratory abnormalities, or other social or family reasons.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: D2 gastrectomy followed by R0 resection, and postoperative pathology confirmed stage II-III gastric cancer
Sampling Method: Probability Sample
Enrollment: 197 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-Free Survival (DFS) rate | 3-year after the last subject participating in
  The 3-year DFS rate is defined as the percentage of patients who remain free of tumor recurrence or death within three years after surgery.

SECONDARY OUTCOMES:
Rate of De-escalation Treatment | 3-year after the last subject participating in
  The Rate of De-escalation Treatment is defined as the proportion of patients among a study population who receive a reduction in the intensity or scope of therapeutic interventions.
Disease-Free Survival (DFS) | 3-year after the last subject participating in
  Disease-Free Survival (DFS) is defined as the duration of time from the initiation of surgery until the recurrence of the disease or death from any cause, whichever comes first.
Cumulative Risk of Recurrence | 3-year after the last subject participating in
  The Cumulative Risk of Recurrence is defined as the cumulative probability or risk of disease recurrence over a specified period, considering the entire study population.
3-year Overall Survival (OS) Rate | 3-year after the last subject participating in
  3-year Overall Survival (OS) Rate is defined as the percentage of patients who are still alive three years after the initiation of a specific treatment, regardless of disease recurrence or progression.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Qilu Hospital of Shandong Univertisy, Jinan, Shandong
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Jinan Central Hospital,, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong

IPD SHARING:
Plan to Share IPD: No